CLINICAL TRIAL: NCT05447832
Title: Remote Monitoring to Predict and Prevent Asthma Attacks in Preschool Children
Brief Title: Remote Monitoring in Preschool Wheeze
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Collaborators: Engineering and Physical Sciences Research Council, UK (Other)
Responsible Party: Principal Investigator, Sejal Saglani, Professor, Imperial College London
Other Study IDs: 307300
Record Dates: First submitted 2022-06-23; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Wheezing; Respiratory Sounds
Keywords: Preschool Wheeze; Asthma Attack
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/Children aged between 1-5 years from the emergency department: Children who have attended the emergency department at St Mary's Hospital, with an acute attack of wheezing. These families will be asked to use the lung function monitoring and the wheeze detection device every night for 2 weeks, while recording symptoms and medication use in the last 24 hours.
  Interventions: Device: Lung function monitoring equipment at home - 2 weeks
- 2/Children aged between 1-5 years admitted electively for wheezing investigation: Children who have been admitted electively for investigations of their wheezing at the Brompton Hospital. These children/families will be asked to do the lung function monitoring and the wheeze detection device once per week for 4 months, while recording symptoms and medication use in the last 24 hours.
  Interventions: Device: Lung function monitoring equipment at home - 4 months; Diagnostic Test: Inflammation and remodelling from clinical indicted bronchoscopy

INTERVENTIONS:
Device: Lung function monitoring equipment at home - 2 weeks — The parent/carer setup the lung function monitoring equipment (Ventica®), and placed the WheezeScan® device on the child's chest at home before the child goes to sleep. This is performed once daily for 2 weeks.
  Groups: 1/Children aged between 1-5 years from the emergency department
Device: Lung function monitoring equipment at home - 4 months — The parent/carer setup the lung function monitoring equipment (Ventica®), and placed the WheezeScan® device on the child's chest at home before the child goes to sleep. This is performed once weekly for 4 months.
  Groups: 2/Children aged between 1-5 years admitted electively for wheezing investigation
Diagnostic Test: Inflammation and remodelling from clinical indicted bronchoscopy — For patients who are undergoing clinically indicated bronchoscopy, consent will be obtained to use any surplus clinical samples for this study. The samples to be collected are broncho-alveolar lavage and endobronchial biopsies. Both of these are taken from the airways during clinical bronchoscopy.
  Groups: 2/Children aged between 1-5 years admitted electively for wheezing investigation

SUMMARY:
The aim of this project is to fill the significant unmet healthcare need to prevent wheeze attacks in preschool children. This will be achieved by developing a proof-of-concept, bespoke home remote objective monitoring system for preschool children that can identify early signs before a wheeze attack to allow early intervention and prevention. This study aims to develop methods for recognising child-specific abnormal patterns in time-course lung function data, and wheeze onset providing early warning of deterioration. The prototype system is targeted for use by caregivers of preschool children with wheeze, and will integrate the individual child's information about symptoms, medication use and lung function to alert parents to seek healthcare advice to prevent hospitalisation.

DETAILED DESCRIPTION:
Asthma is the most common childhood non-infectious lung disease in the United Kingdom, affecting ~8% of children. Asthma symptoms include wheezing (a high-pitched whistling sound created by turbulent airflow through narrowed airways) associated with difficulty in breathing and shortness of breath, often with a dry cough. Asthma is characterised by episodic (wheeze attacks) and variable symptoms which fluctuate day-to-day. An asthma, or wheeze attack, is a sudden worsening of symptoms, associated with airway obstruction that requires treatment to open up the airways.

Preschool children (aged 1-5 years) account for the majority (75%) of hospital admissions for acute attacks of wheezing in the UK. Up to half of all preschool children will suffer at least one episode of wheezing by their 6th birthday, and 7.8% of preschool children came to primary care with acute wheezing in 2017 in the UK. Frequent severe wheeze attacks in preschool age are the strongest risk factor for diminished lung function at physiological peak in early adulthood and are associated with chronic obstructive pulmonary disease (COPD) in the sixth decade of life, as well as early all-cause mortality and cardiovascular and metabolic comorbidities. It is therefore vital to prevent wheeze attacks in preschool children.

Preschool children experience a 5-times higher rate of hospitalisation for acute wheeze attacks compared to school-aged children. This suggests overt symptoms present late, and not soon enough, for early intervention to prevent attacks in preschool children. The number of unscheduled healthcare presentations of acute wheeze attacks has not decreased for the last 2 decades for preschool children, while it has been declining for school-aged children and adults, resulting in a high socioeconomic burden in the UK and worldwide.

Failure to prevent wheeze attacks in preschool children is in part due to the absence of age-specific remote and objective monitoring technology for disease severity. Currently, in this age group, symptoms are diagnosed and monitored by subjective assessments of airway obstruction (narrowing). Evidence that the symptoms improve following treatment with inhaled bronchodilators is used as an indirect indication of the presence of reversible airway obstruction, which is a cardinal feature of asthma. In school-aged children and adults, airway obstruction is monitored objectively with lung function tests such as spirometry. Spirometry can be performed remotely at home to aid telemedicine monitoring in asthma. However, spirometry requires a forced expiratory manoeuvre and cooperation from the patient. It can thus only be reliably performed in children over 5 years old. As a result, diagnosis and monitoring of wheezing/asthma in preschool children depends on parental reports, clinical examination and subjective assessment of symptoms, but no objective measures of airway obstruction.

For this study, time-course lung function data will be obtained using a novel home-based wearable device designed for preschool children that detects airway obstruction whilst the child is asleep (Ventica®). Also, eliciting objective confirmation of wheeze will be obtained by the use of the WheezeScan® device, which detects presence/absence of wheeze when placed on the child's chest. This information will contribute to developing an app that combines symptoms, medication use, and lung function to allow wheeze detection and provide a personalised plan for parents to seek healthcare advice.

STUDY HYPOTHESES

1. A mobile-based system integrating data on remote lung function, symptoms and medication use can be used to predict the development of an acute attack of wheeze in children aged 1-5 years.
2. The dynamic change in lung function reflects underlying airway pathology in severe wheezing

STUDY OBJECTIVES

1. To develop a mobile app system that collects data on lung function, symptoms and medication use, and returns personalised prediction for preschool wheezers, empowering parents to self-manage their child's wheeze/asthma.
2. To quantify airway inflammation and remodelling in endobronchial biopsies and broncho-alveolar lavage from a subgroup of preschool children with severe wheezing and relate pathology to the pattern of airway obstruction detected using the Ventica® system.
3. To develop prediction models that integrate patient-specific abnormal patterns in time-course lung function data, symptoms recorded using with and without WheezeScan®, and rescue medication use, providing early warning of deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-5 years
* Doctor diagnosed and confirmed wheeze
* At least one previous attack of wheeze in the previous year
* Parents/carers with access to a smart phone or computer (to allow data to be entered into the online questionnaire)

Exclusion Criteria:

* Prematurity < 34 weeks gestation
* Need for ventilation in the first seven days after birth
* Known cardiac disease
* Known diagnosis of another respiratory condition (e.g. cystic fibrosis, bronchiectasis)

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1-5 years with recurrent wheezing selected from the hospital emergency department and electively investigations.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-11-29 (Estimated); Study Completion 2024-03-29 (Estimated)

PRIMARY OUTCOMES:
Relation of lung function to symptoms and medication use (Group 1) | 2 weeks
  The lung function measured with the Ventica® system measures tidal breathing variability (non-invasive) in order to assist with the diagnosis and monitoring of asthma or asthmatic symptoms in children aged five years and under. It includes 4 electrodes that are placed under the child's arms - with wires that connect to a small recorder, which is included in a vest that is worn overnight. The presence of wheeze would be detected with the WheezeScan® device, this device needs to be placed on the child's chest for 30-60 seconds and it will confirm if wheezing is present. This will be used by families either when they think their child has symptoms or routinely just prior to the lung function monitoring equipment being used. Both devices include European Conformity (CE) certification and are available for purchase commercially. Symptoms and medication use will be collected using an online secure questionnaire that will be accessible from a computer or a mobile phone.
Relation of lung function to symptoms and medication use (Group 2) | 4 months
  The lung function measured with the Ventica® system measures tidal breathing variability (non-invasive) in order to assist with the diagnosis and monitoring of asthma or asthmatic symptoms in children aged five years and under. It includes 4 electrodes that are placed under the child's arms - with wires that connect to a small recorder, which is included in a vest that is worn overnight. The presence of wheeze would be detected with the WheezeScan® device, this device needs to be placed on the child's chest for 30-60 seconds and it will confirm if wheezing is present. This will be used by families either when they think their child has symptoms or routinely just prior to the lung function monitoring equipment being used. Both devices include European Conformity (CE) certification and are available for purchase commercially. Symptoms and medication use will be collected using an online secure questionnaire that will be accessible from a computer or a mobile phone.
Relation of lung function to airway pathology (Group 2) | 4 months
  Information of patients having a planned bronchoscopy will be collected, to relate airway inflammation and remodelling in bronchial biopsies and broncho-alveolar lavage to the pattern of airway obstruction detected using the Ventica® lung function monitoring system. The endobronchial biopsies will quantify the changes that may cause a child to have wheezing, this includes the amount of mucus, smooth muscle and collagen in the biopsy. The results from these analyses will be related to the lung function measurements, to assess whether specific types of changes in the airway samples relate to specific types of changes in lung function.
Develop a prototype app that combine symptoms, medication use and lung function | 4 months
  The mobile app system will collect data on lung function, symptoms and medication use, and will return personalised predictions for preschool wheezers. The prediction model of attacks and loss of symptom control will be trained using the longitudinal data obtained from the children in the study. Change in lung function, and time to normalisation following treatment for wheezing, will be assessed to understand the time taken for full recovery, and whether persistently abnormal lung function, without overt symptoms, may be an early and sensitive sign for a future attack. The relative contributions of each parameter (symptoms, medication use, wheeze detection, lung function, lower airway inflammation) in determining the accuracy of the model will be assessed to determine the added value of lung function monitoring in predicting individualised patterns of loss of control.

CONTACTS AND LOCATIONS:
Overall Officials: Sejal Saglani, MD, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Royal Brompton and Harefield NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No